CLINICAL TRIAL: NCT01172067
Title: Clinical Impact of Cardiac Resynchronization Therapy on Heart Failure Patients With QuickOpt and Echo Optimization
Brief Title: QuickOpt Chronic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR-09-063-AP-HF
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Heart Failure
Keywords: CRT; heart failure; optimization; Timing cycle optimization methods
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quickopt Group (Experimental): the QuickOpt Group patients will be optimized by QuickOpt(IEGM);
  Interventions: Device: Cardiac Resynchronization Therapy
- Echocardiography group (Active Comparator): the Echo Group patients will be optimized by Echo.
  Interventions: Device: Optimization using echocardiography

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy — Patients will be optimized using QuickOpt (IEGM) algorithm installed on the Merlin device programmer within 2 weeks and 3 and 6 months after device implantation.
  Arms: Quickopt Group
Device: Optimization using echocardiography — Optimization of the AV/PV and VV delays using echocardiography
  Arms: Echocardiography group

SUMMARY:
The purpose of this study is to demonstrate that QuickOpt optimization can be as an alternative method for CRTP/D patients' optimization in clinical practice through the comparison of the improvement differences between the CRTP/D patients with different optimization at 12 months after implantation.The hypothesis is that the Heart Remolding parameter (LVESV) improvement of patients using QuickOpt parameters at 12 months after implant is not inferior (10%) to the patients by Echo optimization。

DETAILED DESCRIPTION:
Clinical studies have demonstrated that the AVTI from QuickOptTM related significantly to the max aorta VTI (AVTI) by Echo, the concordance correlation coefficient (CCC) was so high from 0.96 to 0.99.

But up to now, there are no clinical trials to evaluate mid-long term clinical outcome for CRTP/D patients by QuickOptTM and Echo optimization, this is indeed the main purpose of the study; in addition, the clinical impact, the status of arrhythmia and agents of all the enrolled patients, will be evaluated at 1 year after implant.

ELIGIBILITY:
Inclusion Criteria:

* • Patient meets current CRT-P indications and be implanted with an SJM CRT-P device with V-V timing and a compatible lead system

  * Patient is able to provide written informed consent for study participation

Exclusion Criteria:

* • Patient has limited intrinsic atrial activity (≤ 40 bpm)

  * Patient has persistent or permanent AF
  * Patient has a 2o or 3o heart block
  * Patient's life expectancy is <12 months
  * Patient is <18 years old
  * Patient is pregnant
  * Patient is on IV inotropic agents
  * Patients who are ongoing other devices or agents study
  * Patients with heart transplanted or waiting for heart transplant
  * Patients with Hypertrophic and obstructive cardiomyopathy
  * Patients with severe aortic valve and mitral valve stenosis or regurgitation without replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-05; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quickopt Group | Echocardiography Group
Started | 200 | 200
Completed | 153 | 163
Not Completed | 47 | 37

BASELINE CHARACTERISTICS:
Groups:
- QuickOpt Group: Patients will be optimized using QuickOpt (IEGM) algorithm installed on the Merlin device programmer within 2 weeks and 3 and 6 months after device implantation.
- Total: Total of all reporting groups
Arm/Group | QuickOpt Group | Echocardiography Group | Total
Number analyzed (Participants) | 198 | 194 | 392
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 121 | 133 | 254
  >=65 years | 77 | 61 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.38 (11.77) | 59.21 (11.36) | 60.17 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 54 | 103
  Male | 149 | 140 | 289
Region of Enrollment [Number; unit: participants]
  China | 198 | 194 | 392

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Left Ventricular End Systolic Volume (LVESV) at 12 Months Compared to Baseline
Description: The primary outcome is the percent change in LVESV at 12 months compared to baseline. This outcome measure is assessed through evaluation of echocardiograms at both baseline and 12 months, with a decrease in the percent change in LVESV at 12 months indicating clinical improvement. The percent change in patients with devices optimized with QuickOpt is compared with that of patients with devices optimized using standard echocardiography techniques to determine if one method of optimization results in a greater change in LVESV.
Time Frame: Baseline and12 months
Population: A total of 108 patients in the QuickOpt group and 118 patients in the Echocardiography group had LVESV measurements at both baseline and 12 months to allow comparison of the percent change in LVESV.
Measure: Mean (Standard Deviation); unit: Percent change in LVESV
Arm/Group | QuickOpt Group | Echocardiography Group
Number analyzed (Participants) | 108 | 118
Percent change in LVESV | -24.69 (33.86) | -25.13 (36.06)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Quickopt Group | Echocardiography Group
All-Cause Mortality (participants affected / at risk) | 23/198 | 15/194
Serious Adverse Events (participants affected / at risk) | 28/198 | 19/194
Other Adverse Events (participants affected / at risk) | 6/198 | 6/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quickopt Group (N=198) | Echocardiography Group (N=194)
Death (Cardiac disorders) | 15 (15) | 13 (13) — Death; not related to study devices
Hopitalization (Cardiac disorders) | 3 (3) | 1 (1) — Patient hopitalized then expired; death not related to study devices
Heart Failure Deterioration; Death (Cardiac disorders) | 2 (2) | 0 (0) — Heart failure deteriorated; patient expired; SAE not related to study devices.
Cardiopulmonary arrest, death (Cardiac disorders) | 2 (2) | 0 (0) — Patient sustained cardiopulmonary arrest. Patient expired. The death is not related to study devices.
Junctional rhythm, hypotension (Cardiac disorders) | 1 (1) | 0 (0) — Patient sustained junctional rhythm and low blood pressure. The event was considered related to study device. The pace maker was re-interrogated.
Heart failure deterioration, hospitalization (Cardiac disorders) | 0 (0) | 1 (1) — Heart failure deteriorated. Patient hospitalized. The event is not related to study devices.
Heart failure deterioration, elevated left ventricular pacing threshold (Cardiac disorders) | 1 (1) | 0 (0) — Heart failure deteriorated. Left ventricular pacing threshold increased. The event is not related to study devices.
Heart failure deterioration, myocardial infarction, venous thrombosis, death (Cardiac disorders) | 1 (1) | 0 (0) — Heart failure deteriorated. Patient sustained myocardial infarction and venous thrombosis. Patient expired. The death is not related to study devices.
Heart failure deterioration, phrenic nerve stimulation (Cardiac disorders) | 0 (0) | 1 (1) — Heart failure deteriorated. Patient experienced phrenic nerve stimulation. The event was considered related to study devices.
Myocardial ischemia, staged heart bypass surgery (Cardiac disorders) | 0 (0) | 1 (1) — Patient was diagnosed with myocardial ischemia and underwent staged heart bypass surgery. The event is not related to study devices.
Chest distress, short breaths (Cardiac disorders) | 1 (1) | 0 (0) — Patient stated chest distress and short breaths. Patient was hospitalized. The event is not related to study devices.
Cerebral hemorrhage, death (Vascular disorders) | 0 (0) | 1 (1) — Patient sustained cerebral hemorrhage. Patient expired. The death is not related to study devices.
Haematoma, low right atrial lead sensing (Cardiac disorders) | 0 (0) | 1 (1) — Patient sustained haematoma; the right atrial lead sensing decreased. The event is not related to study devices.
pacemaker pocket ulceration (Cardiac disorders) | 1 (1) | 0 (0) — Pacemaker pocket skin ulceration. The event is not related to study devices.
pacemaker reject (Cardiac disorders) | 1 (1) | 0 (0) — Patient's body rejected pacemaker. The event is not related to study devices.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quickopt Group (N=198) | Echocardiography Group (N=194)
Phrenic nerve stimulation (Cardiac disorders) | 1 (1) | 2 (2) — Patient experience phrenic nerve stimulation. The event is not related to study devices.
Elevated left ventricular pacing threshold (Cardiac disorders) | 2 (2) | 0 (0) — Left ventricular pacing threshold increased.
Coronary sinus dissection (Cardiac disorders) | 1 (1) | 0 (0) — Patient sustained coronary sinus dissection; the event is not related to study devices.
Right ventricular lead dislocation/displacement (Cardiac disorders) | 1 (1) | 0 (0) — Right ventricular lead dislocation/displacement; the event is not related to study devices.
Right atrial lead dislocation/displacement (Cardiac disorders) | 0 (0) | 1 (1) — Right atrial lead dislocation/displacement; the event is not related to study devices.
Left ventricular lead dislocation/displacement (Cardiac disorders) | 1 (1) | 0 (0) — Left ventricular lead dislocation/displacement; the event is related to study devices.
Elevated pacing threshold of left ventricular lead; lead dislocation/displacem (Cardiac disorders) | 0 (0) | 1 (1) — Elevated pacing threshold of left ventricular lead; lead dislocation/displacem; the event is related to study devices.
Infection at pacing system (Infections and infestations) | 0 (0) | 1 (1) — Patient sustain infection at pacing system; the event is not related to study devices.
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) — Patient experienced anaphylactic shock; the event is not related to study devices.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes